CLINICAL TRIAL: NCT04481269
Title: A Prospective Randomized Controlled Study on the Clinical Efficacy of a New Surface Modified Composite Coating Orthopedic Implant Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200718
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Open Fractures, Degenerative Osteoarthritis and Degenerative Spinal Diseases
MeSH Terms: conditions — Fractures, Open; Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research Group (Experimental): Research group uses surface-modified composite coated orthopedic implants
  Interventions: Device: Surface-modified composite coated orthopedic implants
- Controls Group (Active Comparator): Controls group uses conventional orthopedic implants
  Interventions: Device: conventional orthopedic implants

INTERVENTIONS:
Device: Surface-modified composite coated orthopedic implants — The surface-modified composite coated orthopedic implants have the capacity of high binding strength, high tissue-inducing activity and intelligent bacteria-resistance. The implant devices are expected to be used in the prevention and treatment of plant-related infections in orthopedic surgeries.
  Arms: Research Group
Device: conventional orthopedic implants — conventional orthopedic implants
  Arms: Controls Group

SUMMARY:
This study is a prospective, randomized, controlled, double-arm, non-inferiority study that will be carried out in China. It aims to compare two implant systems (the research group uses surface-modified composite coated orthopedic implants, and controls group using conventional orthopedic implants) safety and effectiveness. A total of 240 patients were recruited. The recruited patients are randomly divided into groups at a ratio of 1:1 to ensure that the distribution of patients in the treatment group and the control group is consistent. Patients will receive clinical follow-up in the 1, 3, 6, 9 and 12 months postoperatively. The main indicator for evaluation is the postoperative infection rate, and the secondary indicators include the SF-12 scoring scale, EQ-5D patient questionnaire score, fracture healing, malunion, nonunion incidence in the 12th month after surgery, and skin and soft tissue complications Symptom incidence rate. The follow-up data will be used to determine the main safety and effectiveness of the new surface modified composite coated orthopedic implant system.

ELIGIBILITY:
Inclusion Criteria:

* Limb fracture group criteria

  1. Age 18-75 years old, no gender limit
  2. The preoperative diagnosis is clearly Anderson-Gustilo type III open fracture patient
  3. Postoperative diagnosis stage is IIIA or IIIB patients with open fracture
  4. The subject understands the meaning of this project, volunteers to be the subject, and signs to be informed consent
* Joint replacement group criteria

  1. Age 40-75 years old, no gender limit
  2. The patient is clearly diagnosed as degenerative osteoarthritis before the operation, and the postoperative diagnosis is the same as before the operation
  3. Patients can tolerate implantation operation
  4. The subject understands the meaning of this project, volunteers to be the subject, and signs to be informed consent
* Spine patients group criteria

  1. Age 40-75 years old, no gender limit
  2. Before surgery, it is clearly diagnosed as degenerative spine disease and spine requiring intervertebral fusion
  3. Patients can tolerate implantation operation
  4. The subject understands the meaning of this project, volunteers to be the subject, and signs to be informed consent

Exclusion Criteria:

* 1. The subject is pregnant or breastfeeding, or a woman of childbearing age does not agree to take effective contraceptive measures during the period 2. Closed fractures or pathological fractures (such as primary or metastatic tumors) 3. Patients with symptoms of compartment syndrome 4. According to Gustilo-Anderson classification of open fractures into type I and type II patients 5. Multiple injuries, determined by the researcher to be unsuitable for research 6. The patient is allergic to metal plants 7. Combined with certain medical diseases, it is determined by the investigator to be unsuitable for the study, for example metabolic bone disease, sequelae of polio, poor bone quality, poor bone healing 8. The patient has participated in other clinical trials in the past 3 months 9. The patient has contraindications to anesthesia and surgery 10. Patients with congenital malformations, local or systemic infections, skin diseases 11. The patient is currently receiving chemotherapy or radiotherapy, systemic corticosteroid, long-term use of sedative and hypnotics (using more than 3 consecutive months) or non-steroidal anti-inflammatory drugs (continuous use for more than 3 months) 12. The patient's compliance is poor, and the research staff determines that it cannot be completed according to the research plan. No consent for voluntary participation in clinical research was provided.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
post-operation infection rate | 12 months

SECONDARY OUTCOMES:
SF-12 score | 12 months
EQ-5D score | 12 months
fracture union, malunion, nonunion rate | 12 months